CLINICAL TRIAL: NCT07070193
Title: Retrospective and Prospective Longitudinal Observational Study on Immune Thrombocytopenia Complicated With Acute Ischemic Stroke
Brief Title: Longitudinal Cohort Study on Immune Thrombocytopenia Complicated With Acute Ischemic Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Jiangsu province hospital of TCM (Unknown); Army Medical University, China (Other); Henan Cancer Hospital (Other Government); Ningbo University Affiliated People's Hospital (Unknown); West China Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Zhejiang University (Other); The Second Hospital Of Hebe Medical University (Unknown); Kunming Medical University Second Affiliated Hospital (Unknown); Shanghai Zhongshan Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Huazhong Science & Technology Shanxi Baiqiu En Hospital (Unknown); NORTHERN JIANGSU PEOPLE'S HOSPITAL 1900 (Unknown); Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology (Unknown); Xuzhou Medical University Affiliated Hospital of Huaian (Unknown); Affiliated Hospital of Fujian Medical University, Xiehe Branch (Unknown); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First Affiliated Hospital of Guangxi Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Second Xiangya Hospital of Central South University (Other); Xiangya Hospital of Central South University (Other); Qilu Hospital of Shandong University (Other); Southern Medical University - Southern Hospital (Unknown); The Second Hospital of Hebei Medical University (Other); The First Hospital Affiliated to University of Science and Technology of China (Unknown); The First Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); North China University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice President of Peking University Institute of Hematology Affiliation: Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: ITP-AIS2025
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia (ITP); Acute Ischemic Stroke
Keywords: Immune Thrombocytopenia; Acute Ischemic Stroke
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective cohort: Patients whose first visit to our institution and the termination of follow-up both occurred before the opening of this study will contribute to the retrospective cohort.
- Prospective cohort: Patients whose first visit to our institution occur after the opening of this study will contribute to the prospective cohort.
- Retrospective/Prospective cohort: Patients whose first visit to our institution occurred before the opening of this study and whose follow-up will terminate after the opening of this study will contribute to the ambispective cohort.

SUMMARY:
Immune thrombocytopenia (ITP) is an acquired bleeding disorder mediated by immune-related platelet destruction and impaired platelet production. Immune thrombocytopenia may increase the risk of cerebral infarction and represents a relatively uncommon etiology of acute ischemic stroke. This disease is associated with high disability and mortality rates, poses significant therapeutic challenges, and constitutes a serious threat to human health. Therefore, research on the diagnosis, treatment, and prognosis of ITP combined with acute ischemic stroke is of great significance for improving patients' quality of life and survival outcomes. However, most current hematologic cohort studies are based on single-center or limited multicenter sample sizes, lacking comprehensive and large-scale prospective cohort studies. Our center plans to conduct a large-sample, combined retrospective and prospective longitudinal cohort study. This study will register patients' basic information and diagnosis, follow up with patients through questionnaires, telephone calls, video consultations, online platforms, and in-person visits to record treatment and comorbidity data, collect prognostic information, and retrieve hospitalization and outpatient costs through medical record systems. The study aims to provide comprehensive data on the incidence, treatment, prognosis, and healthcare costs of ITP patients with acute ischemic stroke in China.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an immune-mediated acquired bleeding disorder characterized by thrombocytopenia, with normal or increased megakaryocyte counts in the bone marrow but impaired maturation. The estimated incidence in the general population is approximately 2 to 5 cases per 100,000 individuals. The primary clinical manifestation of ITP is bleeding, ranging from mild skin/mucosal bleeding to life-threatening organ hemorrhage. However, some patients also face an increased risk of thrombosis/embolism. Embolic events in critical organs such as the heart and brain can severely impact patients' quality of life and lead to life-threatening complications.

In China, there are approximately 3.94 million new stroke cases annually, of which acute ischemic stroke (AIS) is the most common type, accounting for 69.6% to 72.8% of all new stroke cases. From an epidemiological perspective, AIS is a globally prevalent disease that significantly affects the quality of life and physical health across populations.

Research indicates that immune thrombocytopenia increases the risk of cerebral infarction and represents a relatively uncommon but important etiological factor for acute ischemic stroke. Currently, most cohort studies on ITP in China are either single-center studies or limited multicenter studies with small sample sizes, resulting in insufficient data and a lack of large-scale, longitudinal prospective cohort studies.

This study is a multicenter, retrospective and prospective longitudinal observational study that will enroll patients diagnosed with ITP and concurrent acute ischemic stroke. It will collect baseline patient information and diagnostic data, conduct regular prospective follow-ups via questionnaires, telephone interviews, video consultations, online platforms, and in-person visits, and record treatment regimens, comorbidities, and prognostic outcomes. Additionally, hospitalization and outpatient costs will be extracted from medical records. The study aims to provide comprehensive data on the epidemiology, treatment patterns, clinical outcomes, and healthcare costs of ITP patients with AIS in China, ultimately supporting the development of novel diagnostic and therapeutic strategies and improving long-term bleeding-free survival rates.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with immune thrombocytopenia, and subsequently identified patients with acute ischemic stroke.
2. Since January 1, 2005, patients who received treatment at Peking University People's Hospital.

Exclusion Criteria:

1. For any reason, such as the occurrence of severe mental disorders, the follow-up information may be unavailable;
2. Patients deemed unsuitable for the study by the researchers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed immune thrombocytopenia (ITP) combined with acute ischemic stroke（AIS)
  Diagnostic Criteria for ITP:
  1. Sustained platelet count <100×10⁹/L
  2. Normal or increased megakaryocyte count in bone marrow with maturation defects
  3. Exclusion of other potential causes of thrombocytopenia including: pseudothrombocytopenia, drug-induced thrombocytopenia, viral infections, helicobacter pylori infection, hematologic disorders, autoimmune diseases, hypersplenism, malignancies
  Diagnostic Criteria for AIS:
  1. Acute onset;
  2. Focal neurological deficits (weakness or numbness of one side of the face or limb, language disorders, etc.), with a few cases presenting with comprehensive neurological deficits;
  3. The presence of a responsible lesion on imaging or the symptoms/signs persisting for more than 24 hours;
  4. Elimination of non-vascular causes;
  5. Brain CT/MRI ruling out cerebral hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Prognosis | 5 years
  To analyze the long-term prognosis of patients with immune thrombocytopenia (ITP) combined with acute ischemic stroke, and analyze the risk factors associated with their prognosis.

SECONDARY OUTCOMES:
Overall response rate | 180 days
  To analyze the therapeutic efficacy of patients with ITP with AIS, and analyze the impact factors associated with the efficacy.
Long-term overall remission rate | 1 year
  Proportion of the participants with an overall remission.
Comorbidities | 5 years
  The incidence, risk factors, treatments, and prognosis of complications
Incidence | 5 years
  To describe the incidence of ITP and AIS, and analyze the risk factors associated with these diseases.
Safety of treatment | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Health economic evaluation | 5 years
  To perform hospital stay and hospitalization cost evaluation in patients with thrombosis and hemostasis diseases

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — eking University Institute of Hematology, Peking University People's Hospital